CLINICAL TRIAL: NCT04311047
Title: Preoperative Detection of Lymph Node Metastases in Pancreatic and Periampullary Carcinoma Using Ultrasmall Super Paramagnetic Iron Oxide Nanoparticle Ferumoxtran-10
Brief Title: Preoperative Detection of Lymph Node Metastases in Pancreatic and Periampullary Carcinoma Using USPIO MRI
Acronym: NANO-PANC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We decided to stop inclusions and start analysis after 26 inclusions.
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL52657.091.15; 2015-000822-12 (EudraCT Number)
Record Dates: First submitted 2020-02-26; First posted 2020-03-17 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-03

CONDITIONS: Pancreatic Cancer; Periampullary Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- USPIO-enhanced MRI (Experimental): Ferumoxtran-10 contrast will be intravenously administered 24-36 before performing an MRI scan. The MRI scan will be discussed with the surgeon prior to resection. Findings on MRI will be compared to pathology.
  Interventions: Diagnostic Test: USPIO-enhanced MRI

INTERVENTIONS:
Diagnostic Test: USPIO-enhanced MRI — Administration of USPIO contrast 24-36 hours before MRI scan of the abdomen to detect lymph node metastases.

SUMMARY:
Adenocarcinoma's of the pancreas and periampullary region (distal bile duct, ampulla of Vater and duodenum) are cancers with a poor survival. Good preoperative TNM staging is important to determine the appropriate therapy and prognosis. An important negative prognostic factor is the presence of para-aortic lymph node (LN) metastases which are regarded as distant metastases and precluding a curative resection. Determining LN status, however, is challenging. Ferrotran, (SPL Medical) an ultra-small superparamagnetic iron oxide (USPIO) particle, has proven to be a valuable contrast agent for detecting LN metastases of solid tumours, like prostate and breast cancer, using magnetic resonance imaging (MRI). The aim of this study is to validate USPIO-MRI to pathology in patients with pancreatic or periampullary cancer.

DETAILED DESCRIPTION:
Rationale:

Pancreatic ductal adenocarcinoma (PDA) is a devastating disease with a dismal prognosis which has not improved substantially in the past 40 years. A good preoperative TNM staging is of importance to determine the appropriate therapy and prognosis. An important negative prognostic factor is the presence of para-aortic lymph node metastases which are regarded as distant metastases and therefore precludes a curative resection of the tumor.

In only 33% of cases para-aortic lymph node metastases are detected preoperatively, due to the low sensitivity of CT and conventional MRI. Moreover, after a curative resection in 70% of patients liver metastases or a local recurrence of disease occurs usually in the lymph nodes of the mesenteric root and in the para-aortic lymph nodes. This suggests that at the time of surgery micrometastases in the liver and lymph nodes were already present. Determining lymph node status preoperatively, however, is a challenge. Ferumoxtran-10, an ultrasmall superparamagnetic iron oxide (USPIO) particle has proven to be a valuable contrast agent for detecting lymph node metastases using magnetic resonance imaging (MRI) in various types of cancer (also called nano-MRI). With this study we would like to validate the results of this technique with pathology in patients with pancreatic or periampullary (duodenal, papilla of Vater or distal bile duct) cancer, i.e. in all patients with adenocarcinoma in the pancreatic region. Ultimately improved preoperative staging of pancreatic and periampullary cancer leads to an improved treatment stratification plan. Demonstration of para-aortic lymph nodes could prevent an unnecessary operation with its associated morbidity and mortality and therefore improve quality of life. Additionally, if metastatic lymph nodes are present, it could complement image guided focal therapies on lymph node metastases such as radiotherapy.

Objective:

The first objective is to improve preoperative staging with 3TESLA (3T) NANO-MRI regarding the detection of lymph node metastases in patients with a pancreatic or periampullary adenocarcinoma when compared to a conventional contrast-enhanced CT with histopathology as gold standard. Other objectives are to improve a) the detection of liver metastases, b) the delineation of the tumor and c) the determination of local vessel ingrowth by the tumor. A more fundamentally oriented objective aims to detect "tumor associated macrophages" in a pancreatic carcinoma with an in vivo 3T NANO-MRI.

Study design:

Feasibility study.

Study population:

Patients with a high index of suspicion of pancreatic or periampullary cancer, who are planned for surgery, but will not receive neo-adjuvant radiotherapy.

Intervention:

We will be administering the USPIO contrast agent ferumoxtran-10 and between 24 and 36 hours later will perform a 3 Tesla MRI scan of the patient.

Main study parameters/endpoints:

Sensitivity and specificity both on a nodal level and on a patient level of the 3T MRI scan with USPIO contrast agent for detecting lymph node metastases in pancreatic and periampullary cancer. Sensitivity and specificity both on a lesion level and on a patient level of the 3T MRI scan with USPIO contrast agent for detecting liver metastases in pancreatic cancer. Delineation of the tumor on USPIO-MRI compared to contrast-enhanced CT. Sensitivity and specificity of the 3T MRI scan with USPIO contrast agent regarding ingrowth of tumor into the portomesenteric veins, the superior mesenteric artery and celiac trunc. Detection of tumor associated macrophages in pancreatic or periampullary adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* High index of suspicion of locally resectable or borderline resectable pancreatic or periampullary (= duodenal, papilla of Vater or distal bile duct) cancer
* Signed and dated informed consent

Exclusion Criteria:

* Pregnancy
* Previous pancreatic surgery
* Previous treatment for the pancreatic or periampullary cancer
* Contraindications for 3T MRI
* Contraindications for USPIO based contrast agents (allergy, hereditary hemochromatosis, thalassemia, sickle cell anemia)
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of USPIO MRI on a regional basis | From date of inclusion until date of resection, maximum 30 days.
  Sensitivity and specificity of USPIO-enhanced MRI for the detection of lymph node metastases on a regional basis

SECONDARY OUTCOMES:
Accuracy of USPIO MRI compared to CT | From date of inclusion until date of resection, maximum 30 days.
  Sensitivity and specificity of CT for detection of lymph node metastases.

CONTACTS AND LOCATIONS:
Overall Officials: John John, MD, PhD, Ir, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Litjens G, Nakamoto A, Brosens LAA, Maas MC, Scheenen TWJ, Zamecnik P, van Geenen EJM, Prokop M, van Laarhoven KJHM, Hermans JJ. Ferumoxtran-10-enhanced MRI for pre-operative metastatic lymph node detection in pancreatic, duodenal, or periampullary adenocarcinoma. Eur Radiol. 2024 Dec;34(12):7973-7984. doi: 10.1007/s00330-024-10838-w. Epub 2024 Jun 22. PMID 38907886